CLINICAL TRIAL: NCT04218695
Title: A Pilot Study of the Effect of Prophylactic Antibiotics on Hospitalized Patients With Advanced Cirrhosis
Brief Title: Prophylactic Antibiotics in Admitted Cirrhotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Association for the Study of Liver Diseases (Other)
Responsible Party: Principal Investigator, Zachary Fricker, Instructor, Division of Gastroenterology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020P000050; BIDMC-ABX-pilot-19 (Other: Beth Israel Deaconess Medical Center)
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Results first posted 2022-08-31 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — Ceftriaxone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded placebo-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Experimental): 1 gram intravenous ceftriaxone once daily for up to one week or until end of hospitalization
  Interventions: Drug: Ceftriaxone
- Placebo (Placebo Comparator): Normal saline (50cc) once daily for up to one week or until end of hospitalization
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ceftriaxone — Antibiotic
  Other Names: Rocephin
  Arms: Treatment
Drug: Normal saline — 50cc intravenous once daily
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
In this pilot study, the investigators aim to assess feasibility of subject identification and data collection, including specimen processing, as well as the rate of enrollment for a future, larger study of the effect of empiric antibiotics for all patients with advanced cirrhosis admitted to the hospital without an existing indication for new antibiotic use. Specifically, the investigators will assess the incidence of infection after the time of enrollment and associated outcomes. Subjects will be randomly assigned to receive antibiotics vs placebo.

DETAILED DESCRIPTION:
Cirrhosis is associated with a state of immune-compromise and progressive decompensation, acute on chronic liver failure (ACLF), and death are often caused by bacterial infections. Different sub-groups of patients with cirrhosis at increased risk, i.e. active upper gastrointestinal hemorrhage, low protein ascites, history of spontaneous bacterial peritonitis (SBP), are known to benefit from prophylactic antibiotics. The investigators hypothesize that hospitalized patients with advanced cirrhosis are also at increased risk and thus may benefit from preventive treatment. Subjects will be randomly assigned to receive an antibiotic vs placebo.

ELIGIBILITY:
Inclusion Criteria:

* MELD-Na >= 18
* Cirrhosis as defined by liver biopsy or a composite assessment of available results from imaging, elastography, prior records, and laboratory studies

Exclusion Criteria:

* Inability to obtain consent (from subject or next of kin/legal authorized representative (LAR)
* Allergy to cephalosporins
* Pregnancy (due to limited prospective data regarding safety of ceftriaxone)
* Existing indication for new antibiotics, e.g. upper gastrointestinal hemorrhage or apparent infection
* Use of major immunosuppressive medications (e.g. prednisone 20 mg/day or greater, immunosuppression for solid organ transplant)
* H/o recurrent C difficile infection within the past year (>2) or requiring fecal microbiota transplant (FMT)
* Enrollment in the study protocol during a previous admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary P Fricker, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fricker Z, Jiang G, Patel H, McLaughlin A, Izunza Barba S, Niezen S, Curry M. A randomized study of ceftriaxone for the prevention of infections in hospitalized patients with advanced cirrhosis. Hepatol Commun. 2024 Jan 5;8(1):e0356. doi: 10.1097/HC9.0000000000000356. eCollection 2024 Jan 1. PMID 38180983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled inpatients only. Enrollment proceeded with intermittent interruption due to COVID pandemic.
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 17 | 15
Completed | 16 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [38 to 70] | 62 [44.5 to 79.5] | 59 [38 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 11 | 25
  Other | 2 | 1 | 3
  Unknown | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 2 | 0 | 2
  Non-Hispanic | 13 | 11 | 24
  Unknown | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Infections
Description: Incident bacterial infection after enrollment
Time Frame: For 7 days or until end of hospital stay
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
Participants | 2 | 5

2. Secondary Outcome: Length of Stay
Description: Days in hospital after randomization
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
days | 9 [-5 to 23] | 10 [-2 to 22]

3. Secondary Outcome: Mortality
Description: In-hospital
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
Participants | 1 | 4

4. Secondary Outcome: 30-day Mortality
Description: Includes f/u after discharge
Time Frame: Up to 30-days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
Participants | 2 | 5

5. Other Pre Specified Outcome: Incident C Difficile Colitis
Description: Positive stool toxin/PCR with new onset diarrhea
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
Participants | 0 | 1

6. Other Pre Specified Outcome: Incident ACLF
Description: (by NACSELD) or change in CLIF-C ACLF score
Time Frame: During hospital admission up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
Participants | 5 | 3

7. Other Pre Specified Outcome: Incident Variceal Hemorrhage
Description: Incident variceal hemorrhage
Time Frame: During hospital admission up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
Participants | 0 | 0

8. Other Pre Specified Outcome: Increase in MELD-Na
Description: >2 pts
Time Frame: Upon discharge (or at 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
Participants | 3 | 3

9. Other Pre Specified Outcome: Fungal Infection
Description: Incident fungal infection (by culture data or requirement for new anti-fungal medication)
Time Frame: During hospital admission up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
Participants | 0 | 0

10. Other Pre Specified Outcome: Biomarker of Infection
Description: Procalcitonin
Time Frame: Once at time of randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
ng/mL | 0.25 [0.05 to 0.45] | 0.44 [0.04 to 0.84]

11. Other Pre Specified Outcome: Biomarker of Infection
Description: C-reactive protein
Time Frame: Once at time of randomization
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 17 | 15
mg/L | 9.7 [2.5 to 16.9] | 11.0 [0.9 to 21.1]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 2/17 | 5/15
Serious Adverse Events (participants affected / at risk) | 3/17 | 5/15
Other Adverse Events (participants affected / at risk) | 4/17 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=17) | Placebo (N=15)
Hepatic Failure (Hepatobiliary disorders) | 1 | 2
Cerebral Edema (Hepatobiliary disorders) | 0 | 1
C. diff cile infection (Infections and infestations) | 0 | 1
Decompensated cirrhosis (Hepatobiliary disorders) | 2 | 1
Necrotizing pancreatitis (Gastrointestinal disorders) | 0 | 1
Pseudoaneurysm sma (Vascular disorders) | 0 | 1
Rectus sheath hematoma (Vascular disorders) | 1 | 0
Hospital acquired pneumonia (Infections and infestations) | 0 | 1
Hypotension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=17) | Placebo (N=15)
Nausea (Gastrointestinal disorders) | 1 | 0
Pruritus with rash (Skin and subcutaneous tissue disorders) | 1 | 0
Possible gastrointestinal bleed (Gastrointestinal disorders) | 1 | 0
hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
ventricular tachycardia (Cardiac disorders) | 0 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
UTI (Infections and infestations) | 1 | 0
Hepatic Encephalopathy (Hepatobiliary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT04218695/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT04218695/ICF_001.pdf